CLINICAL TRIAL: NCT00606255
Title: Compliance of Antihypertensive Treatment Study
Brief Title: Compliance of Antihypertensive Treatment Study (CAT Study)
Acronym: CAT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Sang Hong Baek MD,PhD/ Professor of Medicine, KangNam St.Mary's Hospital The Catholic University of Korea
Other Study IDs: CVAL489AKR19T
Record Dates: First submitted 2008-01-28; First posted 2008-02-01 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Hypertension
Keywords: blood pressure; compliance; treatment
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A: Active training group: Electronic Pill-Boxes with SMS service 1/week, training material provided
- B: Passive training group: Electronic Pill-Boxes ,Training material provided
- C: Usual treatment group: Electronic Pill-Boxes, maintain current treatment method

SUMMARY:
Study Rational:

In general, chronic disease without symptoms such as hypertension, the treatment compliance is relative low and is difficult to increase. The low compliance is related to poor prognosis. There are many factors that effect to compliance of antihypertensive drug. Education is one factor that can be controlled by doctors. Therefore, in this study, the compliance of the patients in 3 groups of active training group, passive training group, and no training group (usual treatment group) will be compared to evaluate the effect of training for controlling of hypertension.

DETAILED DESCRIPTION:
Objectives:

Primary objective - The compliance of each group for the antihypertensive drug is evaluated and compared.

The patients are allocated to three groups; active training group, passive training group, no training group (usual treatment group) and training is performed as described below.

* Active training group: Electronic Pill-Boxes with SMS service 1/week, training material provided
* Passive training group: Electronic Pill-Boxes ,Training material provided
* Usual treatment group: Electronic Pill-Boxes, maintain current treatment method

Secondary objective -

* Evaluate other factor that has effect on the compliance of antihypertensive drug.
* Evaluate the blood pressure lowering effect according to the compliance of antihypertensive drug.
* Evaluate the percentage of missed doses, the percentage of delayed doses, the percentage of multiple doses.
* Evaluate the effect of education on the compliance of antihypertensive drug.

Timelines FPFV : Jan, 2008 LPLV: Dec. 2008

Methodology:

This clinical trial is multi center, prospective, randomized, open, observational study.

This study is to compare the compliance for antihypertensive drugs according to different method of patient training and the observation period per patient is 6 month. There is no fixed visit date and the visits are made according to patient's periodic treatment schedules.

To come up with representative and reliable nation wide statistical data, from hospitals nation wide patient who receive drugs (ACE-I, ARB, β-Blocker, CCB, Diuretic) for blood pressure lowering purpose according to the prescription patterns of investigator will be registered.

Number of centers & patients:

No. of centers: 20 general hospitals No. of patients: 1,062 patients

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed as hypertension.
* Hypertension patients diagnosed and treated but not meeting the target blood pressure. (Target blood pressure: SBP<140mmHg and DBP<90mmHg. In case having concomitant disease JNC-VII guideline is followed)
* Patients age over 18

Exclusion Criteria:

* Patients with severe chronic disease
* Patients scheduled for operation within 6 month period.
* Patients currently participating in other clinical study.
* Pregnant, nursing patient and patient with potential to be pregnant.
* Patient who can not or has no intension to participate in compliance check.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ① Patient diagnosed as hypertension.
  ② Hypertension patients diagnosed and treated but not meeting the target blood pressure. (Target blood pressure: SBP<140mmHg and DBP<90mmHg. In case having concomitant disease JNC-VII guideline is followed)
Sampling Method: Probability Sample
Enrollment: 1062 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of missed doses, delayed doses, the percentage of correct dosing period and blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hong Baek, MD, PhD, Principal Investigator — KangNam St.Mary's Hospital The Catholic University of Korea